CLINICAL TRIAL: NCT02923505
Title: Effect of Positive Airway Pressure Therapy on Hospitalization and Mortality in SDB Patients With Comorbid Chronic Obstructive Pulmonary Disease (COPD) or/and Heart Failure (HF)
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Collaborators: Philips Respironics (Industry)
Responsible Party: Sponsor
Other Study IDs: WI_COPD+HF+SDB_16-250
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Sleep-Disordered Breathing; Pulmonary Disease, Chronic Obstructive; Heart Failure
MeSH Terms: conditions — Sleep Apnea Syndromes; Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- SDB+COPD: Patients with sleep-disordered breathing and concomitant chronic obstructive pulmonary disease
  Interventions: Procedure: polygraphy or polysomnography
- SDB+HF: Patients with sleep-disordered breathing and concomitant heart failure
  Interventions: Procedure: polygraphy or polysomnography
- SDB+COPD+HF: Patients with sleep-disordered breathing and concomitant chronic obstructive pulmonary disease and heart failure
  Interventions: Procedure: polygraphy or polysomnography

INTERVENTIONS:
Procedure: polygraphy or polysomnography

SUMMARY:
The aim of the study is to test the hypothesis that treatment of sleep disordered breathing (SDB) in patients with comorbid chronic obstructive pulmonary disease (COPD) and/or heart failure (HF) with positive airway pressure (PAP) is associated with reduced risk for hospitalizations and death, lower health care utilization, and greater cost-effectiveness.

DETAILED DESCRIPTION:
In this retrospective analysis the health care utilization in patients with COPD and HF will be quantified. Data of patients who additionally underwent a polysomnography or polygraphy between 2012 and 2015 are taken into consideration. The data (risk for hospitalization and death, comorbidities, diagnosis and therapy of SDB, costs of health care utilization) will be collected 12 months before and 12 months after diagnosis of SDB.

The patients' medical records will also be reviewed for compliance to treatment for SDB, and the patients will be classified as treated or untreated. The treated group will be divided into two subgroups: those with "good adherence" to PAP therapy (≥ 4 hours PAP use per night) and those with "poor adherence" to PAP therapy (< 4 hours PAP use per night). Healthcare Utilizations, HF or COPD exacerbations and mortality will be identified by reviewing medical records, National database when available, or self-reported by patient or patient's family through phone interview or questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* subjects between 21 to 75 years;
* consecutive patients who underwent polysomnography or polygraphy during the period of 01/01/2012 to 31/12/2015.
* diagnosis of COPD and/or HF

Exclusion Criteria:

* age <21 or >75 years

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient from primary care clinics and sleep medicine centers
Sampling Method: Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
All-cause Healthcare Costs | 2 years
Diagnosis-related Healthcare Costs | 2 years
Adherence to PAP therapy, (% days with usage >=4h/night) | 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- Danish Center for Sleep Medicine, Glostrup Municipality, Denmark
- Centre Hospitalier Universitaire Grenoble Alpes, Pole Thorax et Vaisseaux (PTV), Clinique de Physiologie Sommeil et Exercice, Grenoble, France
- Germany (3):
  - Interdisziplinäres Schlafmedizinisches Zentrum, Charité Universitätsmedizin Berlin, Berlin
  - Schlafmedizinisches Zentrum der Klinik und Polyklinik für Innere Medizin II, Pneumologie, Universitätsklinikum Regensburg, Regensburg
  - Wissenschaftliches Institut Bethanien für Pneumologie e.V., Solingen

IPD SHARING:
Plan to Share IPD: No